CLINICAL TRIAL: NCT03752671
Title: Efficacy and Safety of the Inter-laminar Device IntraSPINE® Associated with Discectomy in the Treatment of Lumbar Disc Herniation. a Single-blind, Randomised, Comparative, Multicentre Clinical Trial Vs. Discectomy Alone.
Brief Title: Efficacy and Safety of IntraSPINE® Associated with Discectomy in the Treatment of Lumbar Disc Herniation.
Acronym: INTREUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Medical (Industry)
Collaborators: Cousin Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2834_INTRASPINE_EC-EUROPE_16
Record Dates: First submitted 2018-11-16; First posted 2018-11-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Disk Herniated Lumbar
MeSH Terms: interventions — Diskectomy

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will be blinded to the randomisation arm. As the procedure is conducted under general anaesthesia, the patient will not be informed whether the procedure which was performed on him/her did or did not result in the implantation of the IntraSPINE® device (which is not visible on radiographs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the IntraSPINE® device associated with discectomy (Experimental)
  Interventions: Device: Insertion of INTRASPINE device; Procedure: Discectomy
- discectomy alone (Active Comparator)
  Interventions: Procedure: Discectomy

INTERVENTIONS:
Device: Insertion of INTRASPINE device — The surgical technique for excision of the disc hernia is the surgeon's usual technique: patient positioning (lying on his/her back or front or in the knee to chest position) the approach to the lumbar disc hernia (interlaminar or interspinous), closure and drainage of the operation site are performed by the surgeon's usual practice.
  IntraSPINE® is positioned once surgery for the disc hernia has been performed. The implant bed is prepared with the assistance of the distractor provided. The choice of implant size is made after positioning the trial device corresponding to the anatomical bed. Once the size has been established the corresponding implant is placed in a cup of physiological saline prior to implantation. Implantation is performed using the appropriate implant holder.
  Arms: the IntraSPINE® device associated with discectomy
Procedure: Discectomy — The surgical technique for excision of the disc hernia is the surgeon's usual technique: patient positioning (lying prone or supine or in the knee to chest position). The approach to the lumbar disc hernia (interlaminar or interspinous), closure and drainage of the operation site are performed using the surgeon's normal practice.
  Other Names: Discectomy without insertion of INTRASPINE device

SUMMARY:
IntraSPINE® is a novel device that, unlike interspinous positioned implants, is unique in being placed more anteriorly in an interlaminar position, closer to the normal center of rotation of the motion segment. Mechanical advantages are thus conferred over more posteriorly positioned devices through the possibility of more physiological 'rocking' type movements in flexion and extension . This enables IntraSPINE® to off-load the facet joints in extension without blocking movement. Having a more anteriorly placed fulcrum also helps control excessive flexion movements by virtue of an improved lever arm in conjunction with an intact posterior tension band.

The underlying hypothesis of this work is that a clinical gain is achieved by adding an IntraSPINE® interlaminar device to discectomy in patients suffering from a lumbar disc herniation. This should result in an improvement in incapacity level and a reduction in pain.

ELIGIBILITY:
Inclusion Criteria:

Disease-related criteria:

* single segment L4-L5 or L5-S1 lumbar disc hernia identified on imaging (lumbar spine MRI)
* median or posterolateral disc hernia.
* failure of correct medical treatment which has not provided lasting symptom relief absence of contraindications to surgical discectomy and implantation of the IntraSPINE®.

Population related criteria:

* subjects of either sex and over 18 years old
* who have given their free informed signed consent to participate in the study
* patients who are able to respond to the questionnaires and who can communicate in the language of the study country
* and who are affiliated to a social security system or have rights from a social security system.

Exclusion Criteria:

Disease-related criteria:

* recurrent disc hernia post-discectomy at any level
* foraminal and extra-foraminal disc hernia
* paralysing disc hernia (score of 3/5 or less) and cauda equina syndrome
* any grade of spondylolisthesis
* degenerative scoliosis ≥ 15°
* osteoporosis or Paget's disease
* BMI > 30
* procedure required on more than one vertebral level
* endoscopic microdiscectomy prohibiting insertion of the IntraSPINE®
* chronic infection
* systemic or metabolic disorders
* active ongoing malignant disease (liable to prevent the study being conducted and does not carry a risk of vertebral lysis)
* occupational disorder responsible for the disease Treatment or device-related criteria
* allergy to any of the constituents of the medical device

Population-related criteria:

* past history of spinal procedure.
* withdrawal of consent
* pregnant women
* breast-feeding women
* participation in a clinical study within 3 months before the initial visit.
* drug addiction
* predictable lack of availability during the study. Patients deprived of their freedom or under legal guardianship.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 12 months of the degree of functional disability associated with lumbar pain will be measured using the Oswestry Disability Index | Baseline and 12 months
  The Oswestry questionnaire provides an assessment of the symptoms and severity of the back pain and repercussions on activities of daily living. The questionnaire contains 10 questions concerning: pain, personal care, carrying loads, walking, seated position, standing position, sleep, sex life, social life and travel. Each question offers six answers with a score of 0 to 6 which the patient must select: a score of 0 represents normal function and a score of 6 represents greatly reduced function.
  The score obtained is multiplied by 2 in order to obtain a percentage handicap, with 0% for no handicap and 100% for the greatest handicap. It takes approximately 5 minutes to complete the test.

SECONDARY OUTCOMES:
The effect of the IntraSPINE® device associated with discectomy versus discectomy alone in the treatment of lumbar disc herniation with regard to recurrence of disc herniation during the study | All study period (24 months)
  recurrence will be defined as the occurrence of disc herniation confirmed by imaging(MRI) or following surgery at the instrumented level in patients undergoing further surgery during the course of the study. This definition enables the inclusion of all hernias (both symptomatic and asymptomatic).
Evolution between inclusion, 1, 6,12 and 24 months post-surgery of the degree of functional disability like symptoms and severity of back pain and repercussions on activities of daily living associated with lumbar pain using the Oswestry Disability Index | inclusion, 1 month, 6 months, 12 months and 24 months post-surgery
  The Oswestry questionnaire provides an assessment of the symptoms and severity of the back pain and repercussions on activities of daily living. The questionnaire contains 10 questions concerning: pain, personal care, carrying loads, walking, seated position, standing position, sleep, sex life, social life and travel. Each question offers six answers with a score of 0 to 6 which the patient must select: a score of 0 represents normal function and a score of 6 represents greatly reduced function.
  The score obtained is multiplied by 2 in order to obtain a percentage handicap, with 0% for no handicap and 100% for the greatest handicap. It takes approximately 5 minutes to complete the test.
  The Oswestry Disability Index will be measured at inclusion and at 1 month, 6 months, 12 months and 24 months after surgery.
Evolution between inclusion, 1 month, 6 months, 12 months and 24 months post-surgery in the two groups with regard to lumbar and radicular pain using a Visual Analogic Scale | inclusion, 1 month, 6 months, 12 months and 24 months post-surgery
  Radicular and lumbar pain will be assessed on a Visual Analogic Scale at inclusion, 1 month, 6 months, 12 months and 24 months post-surgery. The visual analogue scale is a graduated ruler from 0 to 10 cm where 0 indicates that the subject has no pain and 10 cm represents the maximum pain the subject can tolerate. It is a self-assessment scale and is sensitive, reproducible, reliable and validated both in acute pain and chronic pain situations.
Evolution between inclusion, 12 months and 24 months post-surgery in the two groups with regard to disc height | inclusion, 12 months and 24 months post-surgery
  Disc height (anterior and posterior) will be measured at inclusion, 12 months and 24 months post-surgery based on full-spine x-rays
Evolution between inclusion, 1month, 6 months, 12 months and 24 months post-surgery in the two groups with regard to quality of life | inclusion, 1 month, 6 months, 12 months and 24 months post-surgery
  Quality of life will be assessed using the 12-Item Short Form Survey (SF-12) score at inclusion, 1 month, 6 months, 12 months and 24 months post-surgery.The SF-12 test is a shortened version of the "Medical Outcomes Study Short-Form General Health Survey" (SF 36) which only includes 12 of the 36 questions. The SF 12 provides two scores: a mental and social quality of life score and a physical quality of life score. The SF-12 summary scores range from 0 to 100 with higher scores representing better self-reported health
Evolution between inclusion, 12 months and 24 months post-surgery in the two groups with regard to sagittal alignement | inclusion, 12 months and 24 months post-surgery
  Sagittal alignment will be measured at inclusion, 12 months and 24 months post-surgery by lateral x-ray (full spine).
Evolution between inclusion, 1 month, 6 months, 12 months and 24 months in the two groups with regard to neurological and motor status | inclusion, 1 month, 6 months, 12 months and 24 months
  Neurological and motor status will be assessed at inclusion, 1 month, 6 months, 12 months and 24 months post-surgery using the AIS scale (ASIA "American Spinal Injury Association" Impairment Scale): the section concerning ponytail syndrome will be included in the evaluation.The AIS measurement scale (ASIA "American Spinal Injury Association" Impairment Scale), based on the Frankel Scale is a scale administered by the clinician used to classify the severity of the lesions of patients who have spinal lesions. It is a 5 point ordinal scale and classifies people from A "complete lesions" to E "normal sensory and motor functions"
Time to resumption of work post-surgery | 1 month, 6 months, 12 months and 24 months post-surgery
  The time to resumption of work following surgery will be evaluated in terms of the number of days between hospitalisation and resumption of activity and by the number of days off work due to the disease for which the operation was performed during the 24-month follow-up period.
Rates of further surgery at the level of the implant during the study | All study period (24 months)
  The revision surgery rate (Re intervention or further surgery) . Further surgery throughout the duration of the study is defined as a second operation at the instrumented level (level of the implant performed ) during the course of the study, regardless of reason (i.e. infectious or mechanical): revision, implant removal (explantation), fusion, need for additional fixation, or any surgery affecting any part of the device or relating to any associated complications
The number of adverse events (AE) reported, classified by type and organ. | All study period (24 months)
  The safety and tolerability end points will be will be as follows:
  The number of adverse events (AE) reported, classified by type and organ.
The number of serious adverse events (SAE) reported, classified by type and organ. | All study period (24 months)
  The safety and tolerability end points will be will be as follows:
  The number of serious adverse events (SAE) reported, classified by type and organ.
Integrity of the implant: migration or wear | All study period (24 months)
  The safety and tolerability end points will be will be as follows:
  Integrity of the implant: migration or wear.
The peroperative complication rate. | All study period (24 months)
  The safety and tolerability end points will be will be as follows:
  The peroperative complication rate.
The short and long term postoperative complication rate. | All study period (24 months)
  The safety and tolerability end points will be will be as follows:
  The short and long term postoperative complication rate.

CONTACTS AND LOCATIONS:
Locations (1):
- George Pompidou European Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae J, Lee SM, Lee SH, Shin SH, Kim HJ, Kim KH. The Likelihood of Reaching Substantial Clinical Benefit After an Interlaminar Dynamic Spacer for Chronic Low Back Pain: A Clinical and Radiologic Analysis of a Prospective Cohort. World Neurosurg. 2017 May;101:589-598. doi: 10.1016/j.wneu.2017.02.083. Epub 2017 Feb 27. PMID 28242487
- [Background] Schmidt S, Franke J, Rauschmann M, Adelt D, Bonsanto MM, Sola S. Prospective, randomized, multicenter study with 2-year follow-up to compare the performance of decompression with and without interlaminar stabilization. J Neurosurg Spine. 2018 Apr;28(4):406-415. doi: 10.3171/2017.11.SPINE17643. Epub 2018 Jan 26. PMID 29372860
- [Background] Galarza M, Gazzeri R, De la Rosa P, Martinez-Lage JF. Microdiscectomy with and without insertion of interspinous device for herniated disc at the L5-S1 level. J Clin Neurosci. 2014 Nov;21(11):1934-9. doi: 10.1016/j.jocn.2014.02.029. Epub 2014 Oct 3. PMID 25288390